CLINICAL TRIAL: NCT06561165
Title: Personalizing Multifocal Transcranial Direct Stimulation Dose to Target the Motor Network in Older Adults
Brief Title: Multifocal HD-tDCS and Motor Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Medical University of South Carolina (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael Vesia, PhD, Assistant Professor of Kinesiology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: HUM00250171; 5P2CHD086844-10 (NIH)
Record Dates: First submitted 2024-08-16; First posted 2024-08-19 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Functional Magnetic Resonance Imaging (fMRI); High-density transcranial direct current stimulation; manual dexterity; Non-invasive brain stimulation
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Participants will be randomized and counterbalanced to arm 1 or arm 2.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- HD-tDCS with standard intervention (Experimental): Participants will have three daily sessions.
  Interventions: Device: Standard HD-tDCS intervention; Device: Functional Magnetic Resonance Imaging (fMRI)
- Personalized dose-controlled multifocal network-targeted HD-tDCS. (Experimental): Participants will have three daily sessions.
  Interventions: Device: Multifocal network targeted HD-tDCS intervention; Device: Functional Magnetic Resonance Imaging (fMRI)

INTERVENTIONS:
Device: Standard HD-tDCS intervention — Participants will have three sessions along with behavioral assessments.
  Arms: HD-tDCS with standard intervention
Device: Multifocal network targeted HD-tDCS intervention — Participants will have three sessions along with behavioral assessments.
  Arms: Personalized dose-controlled multifocal network-targeted HD-tDCS.
Device: Functional Magnetic Resonance Imaging (fMRI) — Participants will have an MRI before or after having HD-tDCS intervention.

SUMMARY:
The purpose of this study is to understand how the brain controls movement and how Non-invasive Brain Stimulation (NIBS) with a technique called High-density transcranial direct current stimulation (HD-tDCS) can alter brain processes to improve behavior. Participants in this study will be randomized to either HD-tDCS with standard intervention or personalized dose-controlled multifocal network-targeted HD-tDCS.

The hypothesis is that dexterous hand function will improve after a standard HD-tDCS dose and increase even more after personalized dose-controlled multifocal network-targeted HD-tDCS.

DETAILED DESCRIPTION:
This project is the first of two projects. The second project will be registered as a separate project in the future and enroll participants from this project.

ELIGIBILITY:
Inclusion Criteria:

* Participants should be in good health with normal or corrected-to-normal visual acuity
* Right handed
* No history of neurological disorder
* English speaker
* Able to provide written consent prior to admission

Exclusion Criteria:

* Left-handed
* Participants are pregnant, suspect pregnancy or are attempting to become pregnant
* Have a pacemaker, intracardiac lines or any other medically implanted device or medicine pump
* Have cochlear hearing implants
* Taking drugs known to influence neural receptors that facilitate neuroplasticity (see protocol)
* Have non removable body piercings or have foreign objects in body
* Have metal anywhere in the head that could increase risk of serious injury (not including braces, dental fillings, etc.) (see protocol)
* Have a personal or family history of seizure/epilepsy
* Taking prescription drugs that lower the threshold for seizures
* Recent history of excessive alcohol consumption
* History of alcohol addiction/dependence
* Recent history of recreational drug use
* History of drug addiction/dependence
* Recent history of recreational drug use
* History of drug addiction/dependence
* Diagnosed with a stroke, brain hemorrhage, brain tumor, encephalitis.
* Diagnosed with multiple sclerosis
* Diagnosed with Parkinson's disease or Alzheimer's disease
* Diagnosed with depression in the past 6 months
* Diagnosed with attention deficit disorder, schizophrenia, manic depressive (bipolar) disorder
* Diagnosed with normal pressure hydrocephalus or increased intra-cranial pressure
* Diabetes requiring insulin treatment
* Any serious heart disorder or liver disease

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Percent change in precision force-tracking task | Baseline and 24 hours after the third sessions are completed
  Squared distance (error) from the cursor to the target in precision force-tracking task, estimated as the root mean squared error (RMSE).
Percentage change in the time to complete the nine-hole peg test (9-HPT) | Baseline and 24 hours after the third sessions are completed
  9-hole peg test is a manual dexterity measure, estimated as the time required to complete the task (seconds).

SECONDARY OUTCOMES:
Percentage change in the mean choice reaction time | Baseline and 24 hours after the third sessions are completed
  Mean reaction time for subjects responding in the 2-choice reaction time control task, for correct responses

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vesia, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No